CLINICAL TRIAL: NCT01079741
Title: Phase I/Phase II Open Label Study of the TLR3 Agonist Poly-ICLC as an Adjuvant for NY-ESO-1 Protein Vaccination With or Without Montanide ® ISA-51 VG in Patients With High Risk Melanoma in Complete Clinical Remission
Brief Title: Safety Study of Adjuvant Vaccine to Treat Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nina Bhardwaj (Other)
Collaborators: Ludwig Institute for Cancer Research (Other); Oncovir, Inc. (Industry); Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Director, Tumor Vaccine Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1391
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-11

CONDITIONS: Melanoma
Keywords: Melanoma; Skin Cancer; Adjuvant Therapy; Oncogenesis; LAGE; Cancer Immunity; Neoplasms; Immunogenicity; Vaccine; Immunotherapy
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Carcinogenesis; Neoplasms | interventions — poly ICLC; Monatide (IMS 3015); Poly I-C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose-escalation component (Experimental): Phase I represents the dose-escalation component with Poly-ICLC given in combination with NY-ESO-1 and Montanide in an open-label fashion. The dose of Poly-ICLC will be increased stepwise from 0.35mg to 1.4mg while the dose of NY-ESO-1 antigen and Montanide will be held constant.
  Interventions: Biological: NY-ESO-1 protein; Poly-ICLC; Montanide
- Phase II is the randomized component. (Active Comparator): The doses of NY-ESO-1 and Montanide will remain the same as in Phase I; the highest tolerated Phase I dose of Poly-ICLC will become the Phase II Poly-ICLC dose. In Phase II, patients will be randomized to a subcutaneous vaccination of NY-ESO-1 protein with Poly-ICLC alone dose TBD (Arm A) or with NY-ESO-1 protein, Poly-ICLC dose TBD and Montanide (Arm B).
  Interventions: Biological: NY-ESO-1 protein; Poly-ICLC; Montanide

INTERVENTIONS:
Biological: NY-ESO-1 protein; Poly-ICLC; Montanide — Phase I represents the dose-escalation component with Poly-ICLC given in combination with NY-ESO-1 and Montanide in an open-label fashion. The dose of Poly-ICLC will be increased stepwise from 0.35mg to 1.4mg while the dose of NY-ESO-1 antigen (100µg) and Montanide (1.1mL) will be held constant.
  Phase II: The doses of NY-ESO-1 and Montanide will remain the same as in Phase I; the highest tolerated Phase I dose of Poly-ICLC will become the Phase II Poly-ICLC dose. In Phase II, patients will be randomized to a subcutaneous vaccination of NY-ESO-1 protein with Poly-ICLC alone dose TBD (Arm A) or with NY-ESO-1 protein, Poly-ICLC dose TBD and Montanide (Arm B).
  Other Names: Cancer-Testis (CT) antigen expression: NY-ESO-1; Poly ICLC: carboxymethylcellulose, polyinosinic-polycytidylic acid & poly-L-lysine double-stranded RNA; Montanide® ISA-51 VG: mineral oil-based adjuvant; also called (IFA)incomplete Freund's adjuvant.

SUMMARY:
The incidence of melanoma is increasing with an estimated incidence of 59,940 cases and an annual death rate of 8110 in 2007. Although patients diagnosed with early stage disease have an excellent clinical outcome, patients diagnosed with advanced or recurrent disease, continue to have a high mortality rate, even with initial optimal surgical resection. Effective adjuvant strategies are needed to increase the time to progression and to decrease the recurrence rate. Immunotherapy has long been recognized as a potential therapy for melanoma; the goal of adjuvant vaccine therapy is to train the endogenous immune system to recognize and target minimal residual disease.

DETAILED DESCRIPTION:
This is a Phase I open label dose escalation study of the TLR3 agonist Poly-ICLC as an adjuvant for NY-ESO-1 protein vaccination in patients with high risk melanoma in clinical complete remission (cCr), followed by a randomized Phase II component in which patients will be randomized to subcutaneous vaccination of NY-ESO-1 protein with Poly-ICLC alone dose TBD (Arm A) or with NY-ESO-1 protein, Poly-ICLC dose TBD and Montanide® ISA-51 VG (Montanide) (Arm B).

Patients with histological confirmed malignant melanoma, AJCC Stages: IIB, IIC, III or IV, who are in complete clinical remission (cCr) but at high risk of disease recurrence, will be eligible for enrollment, regardless of whether antigen expression in the autologous tumor can be demonstrated by either PCR or immunohistochemistry.

Primary Objectives:

* Phase I: To define the safety of subcutaneous vaccination with NY-ESO-1 protein, Montanide and escalating doses of Poly-ICLC.
* Phase II: To evaluate the induction of humoral and T cell (CD4+ and CD8+) immunity to subcutaneous vaccination with NY-ESO-1 protein in combination with Poly-ICLC when given with or without Montanide.

Exploratory analyses:

* Evaluation of primary tumor expression of NY-ESO-1 by IHC or RT-PCR.
* Histologic quantitation of original tumor TILs (tumor infiltrating lymphocytes), CD3+ cells, evaluation of mitotic index and correlation of this data with immunologic response.
* Correlation of NY-ESO-1 specific T cell responses with HLA type
* Investigation of polymorphisms for TLR3 through germline SNP analysis.
* Clinical Outcome (Time to Progression) reported descriptively.
* Skin section analysis of protein/adjuvant treated sites for immune cell infiltration and gene expression analysis

ELIGIBILITY:
Inclusion Criteria

1. Histological diagnosis of malignant melanoma, stages IIB-IV in radiologically confirmed cCr without clinical evidence of disease.
2. At least 4 weeks since surgery prior to first dosing of study agent.
3. Laboratory values within the following limits:

   1. Hemoglobin > 10.0 g/dL
   2. Neutrophil count > 1.5 x l09/L
   3. Lymphocyte count > Lower limit of institutional normal
   4. Platelet count > 80 x l09/L
   5. Serum creatinine < 2.0 mg/dL
   6. Serum bilirubin < 2 x upper limit of institutional normal
   7. AST/ALT < 2 x upper limit of institutional normal
4. Patients must have an ECOG performance status of <2 (ECOG criteria published in [67].
5. Life expectancy > 6 months.
6. Age > 18 years.
7. Able and willing to give written informed consent for participation in the trial (see Section 12.2).

Exclusion Criteria

1. Serious illnesses, e.g., serious infections requiring antibiotics.
2. Previous bone marrow or stem cell transplant.
3. History of immunodeficiency disease (such as HIV) or autoimmune disease except vitiligo.
4. Metastatic disease to the central nervous system.
5. Other malignancy within 3 years prior to entry into the study, except for treated early-stage melanoma or non-melanoma skin cancer, or cervical carcinoma in situ.
6. Prior chemotherapy or vaccine therapy.
7. Radiation therapy, biological therapy or surgery within 4 weeks prior to first dose of study agent.
8. Concomitant treatment with systemic corticosteroids greater than physiologic doses. Topical (but not at the proposed vaccination sites) or inhalational steroids are permitted.
9. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent.
10. Pregnancy or lactation.
11. Women of childbearing potential not using a medically acceptable means of contraception.
12. Psychiatric or addictive disorders that may compromise the ability to give informed consent.
13. Lack of availability of the patient for immunological and clinical follow-up assessment.
14. Children <18 years of age who cannot undergo the leukapheresis procedure, do not meet the disease staging and/or the size criteria for frequent blood donations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03-11 (Actual); Study Completion 2013-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — NYU Langone Health; Anna Pavlick, D.O., Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- See also: Click here for more information about this study: Poly-ICLC as an adjuvant for NY-ESO-1 protein vaccination with or without Montanide ® ISA-51 VG in patients with high risk melanoma in complete clinical remission — http://www.med.nyu.edu/clinicaltrials/

RESULTS

PARTICIPANT FLOW:
Groups:
- Poly-ICLC 0.35mg: Cohort 1 100µg NY-ESO-1 protein + 1.1 mL Montanide + 0.35mg Poly-ICLC. The cycle was repeated every 3 weeks for a total of 4 cycles.
- Poly-ICLC 0.7mg: Cohort 2 100 µg NY-ESO-1 protein + 1.1 mL Montanide + 0.7mg Poly-ICLC.The cycle was repeated every 3 weeks for a total of 4 cycles.
- Poly-ICLC 1.4mg: Cohort 3 100 µg NY-ESO-1 protein + 1.1 mL Montanide + 1.4 mg Poly-ICLC. The cycle was repeated every 3 weeks for a total of 4 cycles.
- NY-ESO-1 Protein and Poly-ICLC: Phase 2, Arm 1 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC.
- NY-ESO-1 Protein, Poly-ICLC and Montanide: Phase 2, Arm 2 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC and 1.1mL Montanide.
Period: Cohort 1: Dose Level 1 (Weeks 1-12)
Arm/Group | Poly-ICLC 0.35mg | Poly-ICLC 0.7mg | Poly-ICLC 1.4mg | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Started | 3 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 2 (Weeks 13-24)
Arm/Group | Poly-ICLC 0.35mg | Poly-ICLC 0.7mg | Poly-ICLC 1.4mg | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Started | 0 | 4 | 0 | 0 | 0
Completed | 0 | 3 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0
Period: Cohort 3: Dose Level 3 (Weeks 25-36)
Arm/Group | Poly-ICLC 0.35mg | Poly-ICLC 0.7mg | Poly-ICLC 1.4mg | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0
Period: Phase 2 (Weeks 37-48)
Arm/Group | Poly-ICLC 0.35mg | Poly-ICLC 0.7mg | Poly-ICLC 1.4mg | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Started | 0 | 0 | 0 | 12 | 12
Completed | 0 | 0 | 0 | 12 | 9
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Poly-ICLC 0.35 mg: Cohort 1 100µg NY-ESO-1 protein + 1.1 mL Montanide + 0.35mg Poly-ICLC. The cycle was repeated every 3 weeks for a total of 4 cycles.
- Poly-ICLC 0.70 mg: 100 µg NY-ESO-1 protein + 1.1 mL Montanide + 0.7mg Poly-ICLC.The cycle was repeated every 3 weeks for a total of 4 cycles.
- Poly-ICLC 1.4mg: 100 µg NY-ESO-1 protein + 1.1 mL Montanide + 1.4 mg Poly-ICLC. The cycle was repeated every 3 weeks for a total of 4 cycles.
- NY-ESO-1 Protein and Poly-ICLC: 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC.
- NY-ESO-1 Protein, Poly-ICLC and Montanide: 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC and 1.1mL Montanide.
- Total: Total of all reporting groups
Arm/Group | Poly-ICLC 0.35 mg | Poly-ICLC 0.70 mg | Poly-ICLC 1.4mg | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide | Total
Number analyzed (Participants) | 3 | 4 | 3 | 12 | 12 | 34
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 72] | 65 [39 to 74] | 73 [64 to 78] | 50 [21 to 69] | 57 [24 to 83] | 55 [21 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 5 | 6 | 13
  Male | 3 | 2 | 3 | 7 | 6 | 21
Pathologic Staging [Count of Participants; unit: Participants] — IIA - Melanoma thickness1-2mm with ulceration or 2-4mm without ulceration; IIB - 2-4 mm thickness with ulceration or 4mm without ulceration IIC - thickness >4mm with ulceration IIIA - thickness any size, no ulcerations, 1-3 nodes micrometasis IIIB - thickness any size, 1-3 nodes, with or without ulcerations, micrometasis or macrometasis IIIC - thickness any size, with or without ulcerations 1-3 nodes, micrometasis, marcrometasis, or in transit mets(s)/satellite(s) without metastatic nodes IV - any thickness, with or without ulcerations, nay nodes, any distant metastases
  Participants
    IIA | 0 | 0 | 0 | 1 | 0 | 1
    IIB | 0 | 0 | 1 | 1 | 0 | 2
    IIC | 1 | 0 | 0 | 0 | 1 | 2
    IIIA | 1 | 0 | 0 | 0 | 2 | 3
    IIIB | 1 | 1 | 0 | 4 | 3 | 9
    IIIC | 0 | 3 | 2 | 4 | 4 | 13
    IV | 0 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase I, Number of Participants With SAE and DLT
Description: Safety measured by number of Serious Adverse Events per the CTEP v4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) and Dose Limiting Toxicity (DLT).
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Poly-ICLC 0.35 mg | Poly-ICLC 0.70 mg | Poly-ICLC 1.4mg
Number analyzed (Participants) | 3 | 3 | 3
Participants
  Serious Adverse Events | 0 | 0 | 1
  DLT | 0 | 0 | 0

2. Secondary Outcome: CD4+ and CD8+ Response
Description: Cellular response evaluated for the induction of cellular T cell (CD4+ and CD8+) immunity to subcutaneous vaccination with NY-ESO-1 protein in combination with Poly-ICLC when given with or without Montanide. Number of participants with increase CD4+ and CD8+ levels.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Number analyzed (Participants) | 12 | 9
Participants
  CD4 Responder | 10 | 9
  CD8 Responder | 1 | 4

3. Secondary Outcome: NY-ESO-1 Expression by IHC
Description: Analysis of immune cell infiltration at the injection site by IHC. IHC analysis of immune cell infiltration was performed for each arm using a scoring system. 0: No expression of the marker of interest, 1: single cells or small clusters (<5 cells together) expressing marker of interest, 2: medium size clusters of cells expressing marker of interest, and 3: huge and homogeneously positive clusters of cells expressing marker of interest.
Time Frame: up to 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NY-ESO-1 Protein and Poly-ICLC | NY-ESO-1 Protein, Poly-ICLC and Montanide
Number analyzed (Participants) | 12 | 9
units on a scale
  CD3 lymphocytes | 1.500 (0.707) | 1.944 (0.682)
  CD4 lymphocytes | 1.318 (0.643) | 2.167 (0.661)
  CD8 lymphocytes | 1.091 (0.437) | 1.222 (0.565)
  CD20 B cells | 0.773 (0.518) | 1.500 (0.500)
  CD11c dendritic cells | 1.455 (0.611) | 2.111 (0.741)

ADVERSE EVENTS:
Groups:
- Phase 2, Arm 1: 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC.
- Phase 2, Arm 2: 100μg NY-ESO-1 protein, 1.4mg Poly-ICLC and 1.1mL Montanide.
Arm/Group | Poly-ICLC 0.35 mg | Poly-ICLC 0.70 mg | Poly-ICLC 1.4mg | Phase 2, Arm 1 | Phase 2, Arm 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 1/3 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poly-ICLC 0.35 mg (N=3) | Poly-ICLC 0.70 mg (N=4) | Poly-ICLC 1.4mg (N=3) | Phase 2, Arm 1 (N=12) | Phase 2, Arm 2 (N=12)
Stent placement (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poly-ICLC 0.35 mg (N=3) | Poly-ICLC 0.70 mg (N=4) | Poly-ICLC 1.4mg (N=3) | Phase 2, Arm 1 (N=12) | Phase 2, Arm 2 (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 2 | 1 | 9 | 8
Injection site erythema (General disorders) | 3 | 3 | 2 | 12 | 9
Injection site nodule (General disorders) | 3 | 3 | 3 | 6 | 12
Injection site edema (General disorders) | 3 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 3 | 3 | 3 | 12 | 12
Fatigue (General disorders) | 2 | 3 | 1 | 10 | 8
Injection site exfoliation (General disorders) | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 6 | 3
Injection site discharge (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 1 | 3 | 2 | 8 | 4
Injection site induration (General disorders) | 1 | 3 | 3 | 0 | 0
Injection site pruritus (General disorders) | 1 | 3 | 1 | 6 | 7
Injection site vesicles (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 5 | 2
Pyrexia (General disorders) | 1 | 1 | 1 | 4 | 4
Injection site urticaria (General disorders) | 0 | 2 | 3 | 0 | 0
Injection site dryness (General disorders) | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Promotion of wound healing (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 6 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 2 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Eye Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 6 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes